

The David Hide Asthma and Allergy Research Centre St Mary's Hospital, Newport, Isle of Wight, PO30 5TG

## **Consent Form**

**Project:** The effect of Dyson Air Purifier in Improving Asthma Control – A Randomised Controlled Trial **Short Title** Dyson Air Purifier in Asthma Researchers: Hasan Arshad Professor and Consultant in Allergy Ramesh Kurukulaaratchy -Consultant in Respiratory Medicine Part A: Please initial boxes 1. I confirm that I have read and understand the information sheet dated \*\*[insert date and version once approved] \*\* for the above study and have had the opportunity to ask questions. 2. I understand that my participation is voluntary and that I am free to withdraw at any time, without giving any reason, and without my medical care or legal rights being affected. 3. I understand that sections of any of my medical notes and/or GP care data may be looked at by members of the research team at the David Hide Asthma and Allergy Research Centre for the purpose of collecting data; and members of the Trust Research Department for audit/monitoring purposes. I give my permission for these individuals to have access to my records. I give permission for my General Practitioner to be informed of my decision to participate in 4. this study and receive the results of my bronchial challenge test(s). 5. I agree to the NHS computer systems being used to confirm contact details now and in the future. 6. I agree to a member of the study team installing 2 Dyson Air Purifiers in my home (1 in the living room and 1 in the bedroom) and I understand that I will not receive any payment as reimbursement of the running costs. I agree to the collection of dust samples from my home. 7. I agree to undertake FeNO measurement and lung function testing including the 8 administration of Methacholine for the study; and to the administration of 400 to 600mcg of salbutamol after the test is complete. 9. I agree to a skin prick test to common aero-allergens. 10. I agree to keep peak flow and symptom diaries according to the study schedule.

Continued over the page...

| 1 for participant, 1 for researcher, 1 to be kept with hospital notes | | | |
|---|---|---|---|
| Nam | e of Person taking Consent | Date | Signature |
| Parti | cipant Name | Date | Signature |
| 3. | . I give permission for a member of the research team to look at my medical records, to obtain information on allergy, asthma and related conditions. I understand that the information will be kept confidential. | | |
| 2. | I give permission for the samples to be used for genetic research aimed at understanding the genetic basis of allergy, asthma and related conditions. | | |
| 1. | I give permission for the samples to be used for investigations of medical conditions relating allergy, asthma and related conditions. | | |
| Part B: Linked anonymised samples gifted for storage and use in future studies: I give permission for samples to be stored (potentially for many years) for possible use in future research studies. Future studies will be reviewed and approved by a Research Ethics Committee prior to the samples being used. I understand that these studies may not directly benefit my health. You can alter these decisions at any stage by letting the researcher know. | | | |
| 18. | I voluntarily agree to participate in the al | oove study. | |
| 17. | behalf of my cohabitants. | | |
| 16. | I give permission for the study team to contact me after the study to discuss further participation in research studies that may be of interest. | | |
| 15. | <ol> <li>I agree to make the Products available for collection when requested by the David Hide<br/>Asthma and Allergy Research Centre</li> </ol> | | |
| 14. | | | |
| 13. | 3. * Female participants only * I agree to provide a urine sample for the purpose of excluding pregnancy prior to performing a Methacholine Challenge. (not applicable if postmenopause) | | |
| 12. | 12. I agree to provide a small sample of blood | | |
| 11. | I agree to complete quality of life questionnaires. | e, environmer | ntal, asthma and rhinitis related |

ı